CLINICAL TRIAL: NCT02561377
Title: Effect of Resistance Training on Metabolic Control and Outcome in Prediabetes (NMR-based Metabonomics)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing University of Traditional Chinese Medicine (Other)
Collaborators: Guangxi Medical University (Other); Southeast University, China (Other)
Responsible Party: Principal Investigator, Lou Qingqing, director, department of education, Nanjing University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 81370923
Record Dates: First submitted 2015-09-24; First posted 2015-09-28 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Prediabetic State
Keywords: resistance training; Prediabetic state; Metabolomics
MeSH Terms: conditions — Prediabetic State | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- resistance training (Experimental): Resistance training consisted of 6 different resistance exercises per session using elastic string, and each exercise progressed to 2-3 at maximum resistance lifted 8-10 times.
  Interventions: Behavioral: resistance training
- aerobic training (Experimental): Aerobic training consisted of aerobic exercise and progressed from 15-20min/session at 60% maximum heart rate to 45-50min/session at 75% maximum heart rate.
  Interventions: Behavioral: aerobic training
- standard care (No Intervention): standard care complied with the daily lifestyle.

INTERVENTIONS:
Behavioral: resistance training — Resistance training consisted of 6 different resistance exercises per session using elastic string, and each exercise progressed to 2-3 at maximum resistance lifted 8-10 times.
  Arms: resistance training
Behavioral: aerobic training — Aerobic training consisted of aerobic exercise and progressed from 15-20min/session at 60% maximum heart rate to 45-50min/session at 75% maximum heart rate.
  Arms: aerobic training

SUMMARY:
This study evaluates the efficacy of a 12-month resistance training on metabolic control and reducing the risk of diabetes.

DETAILED DESCRIPTION:
Most of exercise interventions involved aerobic exercises, investigators were not able to find a single long term study focusing on type 2 diabetes prevention with resistance training and aerobic exercise. It has been known that for those who have already had diabetes, resistance training can reduce insulin resistance and HbA1c level, improve lipid profile, and decrease blood pressure. Based on previous findings, investigators will evaluate how the different exercising interventions impact on insulin resistance, metabolic control, and the incidence and prevalence of diabetes in prediabetes population who receive 12 months of either resistant training or aerobic exercise. Further more, metabolomics approach will be introduced to detect biological markers,and therefore,to analyze the predictive values of metabolomics on long term outcomes of prediabetes population.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of prediabetes according to the American Diabetes Association (ADA) guidelines
* level 4 of muscle strength
* willingness to accept exercise intervention
* provision of written informed consent.

Exclusion Criteria:

* type 2 or other types of diabetes
* women who are pregnant
* hepatic dysfunction, as evidenced by alanine aminotransferase (ALT) or alkaline phosphatase (ALP) levels greater than 2.5-fold the upper limits of normal
* crucial organ failure or other severe diseases, including myocardial infarction
* malignancy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-07 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
glycemic control | 6 months
  Fasting blood glucose, postprandial blood glucose and HbA1c will be measured at 6 months.
glycemic control | 12 months
  Fasting blood glucose, postprandial blood glucose and HbA1c will be measured at 12 months.

SECONDARY OUTCOMES:
small molecule metabolites | 6 months
  Biological markers, with the method of metabolomics approach, will be measured at 6 months
small molecule metabolites | 12 months
  Biological markers, with the method of metabolomics approach, will be measured at 12 months.
Incidence rate of diabetes | 6 months
  Evaluate the incidence of diabetes in prediabetes population at 6 months.
Incidence rate of diabetes | 12 months
  Evaluate the incidence of diabetes in prediabetes population at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Qingqing Lou, Study Director — Nanjing University of Traditional Chinese Medicine
Locations (2):
- China (2):
  - The first Affiliated hospital of Guangxi medical university, Nanning, Guangxi
  - Southeast University, China, Nanjing, Jiangsu

REFERENCES:
- [Background] Morrison F, Shubina M, Turchin A. Lifestyle counseling in routine care and long-term glucose, blood pressure, and cholesterol control in patients with diabetes. Diabetes Care. 2012 Feb;35(2):334-41. doi: 10.2337/dc11-1635. PMID 22275442
- [Background] Lewis GD, Farrell L, Wood MJ, Martinovic M, Arany Z, Rowe GC, Souza A, Cheng S, McCabe EL, Yang E, Shi X, Deo R, Roth FP, Asnani A, Rhee EP, Systrom DM, Semigran MJ, Vasan RS, Carr SA, Wang TJ, Sabatine MS, Clish CB, Gerszten RE. Metabolic signatures of exercise in human plasma. Sci Transl Med. 2010 May 26;2(33):33ra37. doi: 10.1126/scitranslmed.3001006. PMID 20505214
- [Background] Strasser B, Siebert U, Schobersberger W. Resistance training in the treatment of the metabolic syndrome: a systematic review and meta-analysis of the effect of resistance training on metabolic clustering in patients with abnormal glucose metabolism. Sports Med. 2010 May 1;40(5):397-415. doi: 10.2165/11531380-000000000-00000. PMID 20433212
- [Derived] Chen X, Zhao S, Hsue C, Dai X, Liu L, Miller JD, Fang Z, Feng J, Huang Y, Wang X, Lou Q. Effects of aerobic training and resistance training in reducing cardiovascular disease risk for patients with prediabetes: A multi-center randomized controlled trial. Prim Care Diabetes. 2021 Dec;15(6):1063-1070. doi: 10.1016/j.pcd.2021.08.013. Epub 2021 Oct 11. PMID 34649825
- [Derived] Yan J, Dai X, Feng J, Yuan X, Li J, Yang L, Zuo P, Fang Z, Liu C, Hsue C, Zhu J, Miller JD, Lou Q. Effect of 12-Month Resistance Training on Changes in Abdominal Adipose Tissue and Metabolic Variables in Patients with Prediabetes: A Randomized Controlled Trial. J Diabetes Res. 2019 Oct 16;2019:8469739. doi: 10.1155/2019/8469739. eCollection 2019. PMID 31737686